CLINICAL TRIAL: NCT05958563
Title: Impact of Continuous Positive Airway Pressure on the Occurrence of Acute Exacerbations of COPD in Patients With COPD-OSA Overlap Syndrome (CO-OS) SLEEPOVEA
Brief Title: Impact of Continuous Positive Airway Pressure on the Occurrence of Acute Exacerbations of COPD in Patients With COPD-OSA Overlap Syndrome (CO-OS)
Acronym: SLEEPOVEA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49RC21_0377
Record Dates: First submitted 2023-07-12; First posted 2023-07-24 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Sleep Apnea; COPD Exacerbation; Overlap Syndrome
Keywords: sleep apnea; copd; overlap syndrome
MeSH Terms: conditions — Sleep Apnea Syndromes; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: randomized control study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPAP group (Experimental): Continuous positive airway pressure (CPAP) for one year
  Interventions: Device: continuous positive airway pressure treatment
- Control group (No Intervention): No CPAP treatment

INTERVENTIONS:
Device: continuous positive airway pressure treatment — CPAP treatment for one year
  Arms: CPAP group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) and Obstructive Sleep Apnea (OSA) are both frequent respiratory diseases with estimated prevalences between 8 and 15% of the adult population. Because of those high prevalences those two entities are often associated in same patients (1 to 4% of the general population). This association is then referred to as Overlap Syndrome (CO-OS). Data from observational studies suggest that this association may have an additive or even synergistic negative impact on patient's prognosis. Indeed, in a cohort of patients diagnosed as having a CO-OS, patients who did not receive specific treatment for OSA had a 76% increased risk of death compared to patients treated with continuous positive airway pressure (CPAP) and a 2-fold increased risk of acute COPD exacerbation. In another cohort of patients with both OSA and severe oxygen treated COPD, untreated patients for OSA had a 5-fold increased risk of death compared to patients treated with CPAP. There are strong signals from observational studies in support of a beneficial impact of CPAP therapy on respiratory outcomes in patients with CO-OS. However, those findings are not supported by any controlled study. It is difficult to directly transpose the observational data to current clinical practice in the context of the recent studies on the impact of CPAP on OSA prognosis. Indeed, data from similar observational OSA cohorts have reported a major impact of CPAP on the overall survival and cardiovascular outcomes in patients with OSA. Ten years later, this impact has not been confirmed by several randomized studies. To date, there is no consensus on a systematic screening and, if present, management of OSA in patients with COPD. The need for specific research on that field was emphasized in 2018 in an official American Thoracic Society Research Statement which recommends "randomized trials that compare clinical outcomes among patients with Overlap Syndrome whose OSA is treated to clinical outcomes among patients with Overlap Syndrome whose OSA is untreated".

DETAILED DESCRIPTION:
This study is an open labeled parallel group randomized controlled trial. The patients will be recruited within the pneumology consultations of the participating centers. Patients meeting the pre-inclusion criteria and having no exclusion criteria will be included in the study and will undergo a polysomnographic sleep recording (PSG).

Patients with apnea hypopnea index (AHI) <15 / hour and/or significant central apneas (≥5 central apneas per hour of sleep) during PSG will be excluded from the study.

Patients with moderate to severe OSA (AHI ≥15 /h) and no significant central apneas will undergo baseline evaluation (ABG, 6 minute walking test, FEV1 and questionnaires) and then will be randomly assigned to receive 1 year of CPAP treatment (CPAP group) or no treatment of OSA (control group) according to a 1:1 allocation using a computer-generated randomization list stratified by site and OSA severity with permuted blocks of random sizes.

Visit at 3,6 and 9 months: the following outcomes will be assessed: COPD exacerbations (number, date and severity), cardiovascular events, death and questionnaires.

Visit at the end of the study (12 months): the following outcomes will be assessed: COPD exacerbations (number, date and severity), cardiovascular events, death, questionnaires, ABG, 6 minute walking test, FEV1.

Statistical analysis for primary and secondary outcomes will be performed on an intention to treat basis. A per-protocol analysis will be also performed in patients with an average objective CPAP use of at least 4 hours per day. Pre-specified sensitivity analysis will be conducted according to age, gender, body-mass index, OSA and COPD severity.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or older
* Grade of 2 or higher on the modified Medical Research Council scale (which ranges from 0 to 4, with higher grades indicating more severe dyspnea)
* A post-bronchodilator forced expiratory volume in 1 second (FEV1) of less than 70% of the predicted value, and a postbronchodilator ratio of FEV1 to forced vital capacity (FVC) of less than 0.70.
* Documented history of at least one moderate or severe COPD exacerbation during the previous year
* Clinical suspicion of OSA (based on a STOP-bang questionnaire >3),
* Have a telephone or a tablet or accept to use one during the study,
* Willing and able to comply with all study procedures,
* Subjects covered by or having the rights to medical care assurance.
* An apnea-hypopnea index [AHI], ≥15 per hour based on a full night polysomnography and no significant central apneas (<5 central apneas per hour of sleep

Exclusion Criteria:

* Severe daytime sleepiness (Epworth sleepiness Scale >14/24 and/or frequent sleepiness while driving or patient escaping a sleep-onset accident within the last 12 months),
* Severe unstable cardiovascular disease (heart failure with FEVG≤45%, recurrent cardiac arrhythmia, instable coronary heart disease or stroke),
* Patient on long-term oxygen therapy or non-invasive ventilation
* Previously documented severe hypercapnia (PaCO2 ≥ 50mm Hg)
* Previously diagnosed and treated OSA
* Any rehabilitation program or any lung volume reduction procedure planned in the oncoming year
* Pregnancy, breastfeeding
* Bad understanding of the French language,
* Other protected person according to articles L1121.7 and L1121.8 of the French Public Health Act

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
annual rate of COPD exacerbations | 12 months
  COPD exacerbations will be captured using the EXACT-PRO diary. COPD exacerbations will be defined as a worsening of two or more of dyspnea, sputum purulence or sputum volume for at least two consecutive days and captured using an electronic diary (EXACT-PRO) for mild exacerbation or during clinical visits for moderate and severe exacerbations.

SECONDARY OUTCOMES:
Annual rate of moderate to severe COPD exacerbations and severe COPD exacerbations | 12 months
  The type of treatment provided for a COPD exacerbation will determine the severity of the exacerbation. It will be categorized as mild (involving worsening of symptoms for >2 consecutive days), moderate (leading to treatment with glucocorticoids, antibiotics, or both), or severe (leading to hospital admission)
Times to the first COPD exacerbation of any severity | 12 months
  COPD exacerbations will be captured using the EXACT-PRO diary. COPD exacerbations will be defined as a worsening of two or more of dyspnea, sputum purulence or sputum volume for at least two consecutive days and captured using an electronic diary (EXACT-PRO) for mild exacerbation or during clinical visits for moderate and severe exacerbations.
Times to the first COPD exacerbation of the first moderate or severe COPD exacerbation | 12 months
  The type of treatment provided for a COPD exacerbation will determine the severity of the exacerbation. It will be categorized as mild (involving worsening of symptoms for >2 consecutive days), moderate (leading to treatment with glucocorticoids, antibiotics, or both), or severe (leading to hospital admission)
Times to the first COPD exacerbation of the first severe COPD exacerbation | 12 months
  The type of treatment provided for a COPD exacerbation will determine the severity of the exacerbation. It will be categorized as mild (involving worsening of symptoms for >2 consecutive days), moderate (leading to treatment with glucocorticoids, antibiotics, or both), or severe (leading to hospital admission)
Annual rate of non-fatal cardiovascular events | 12 months
  non-fatal myocardial infarction, non-fatal stroke, coronary artery bypass surgery, and percutaneous transluminal coronary angiography
Mortality rate | 12 months
  deaths
Measurement of the quality of life | 12 months
  Saint George's Respiratory Questionnaire
Dyspnea | 12 months
  modified Medical Research Council scale
Functional respiratory | 12 months
  forced expiratory volume in one second
exercise capacity | 12 months
  6 minutes walking test
Daytime sleepiness | 12 months
  Epworth Sleepiness Scale
Subjective sleep quality | 12 months
  Pittsburgh sleep quality index
Arterial blood gases | 12 months
  Partial pressure of oxygen and carbon dioxide

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - Angers University Hospital, Angers
  - Bordeaux University Hospital, Bordeaux
  - Brest University Hospital, Brest
  - AP-HP -Henri Mondor Hsopital, Créteil
  - Dijon University Hospital, Dijon
  - Grenoble University Hospital, Grenoble
  - Le Mans Hospital, Le Mans
  - Nancy University Hospital, Nancy
  - AP-HP - Pitié Salpetrière Hospital, Paris
  - Bichat Hospital - AP-HP, Paris
  - Poitiers University Hospital, Poitiers
  - Reims University Hospital, Reims
  - Polyclinique Saint Laurent, Rennes
  - Strasbourg University Hospital, Strasbourg
  - Toulouse Universty Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided